CLINICAL TRIAL: NCT07043647
Title: A Randomized Controlled Trial of an Agricultural Livelihood Intervention to Improve Maternal and Newborn Health and Nutrition in Kenya: Mama Shamba
Brief Title: An Agricultural Livelihood Intervention for Pregnant Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Kenya Medical Research Institute (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01HD116651 (NIH); R01HD116651 (NIH)
Record Dates: First submitted 2025-06-20; First posted 2025-06-29 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Food Insecurity; Pregnancy; Birth Outcomes; Livelihood Interventions; Infant Health Outcomes
Keywords: Food Insecurity; Pregnancy; Birth Outcomes; Livelihood interventions; agricultural Interventions; Kenya

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Agricultural tools and training (Experimental): Provision of water pump, other supplies, training, and harvest from the demonstration farm in early pregnancy
  Interventions: Other: Shamba Maisha
- Control Arm (No Intervention): Control participants will be offered the full intervention at the conclusion of study follow-up.

INTERVENTIONS:
Other: Shamba Maisha — The Shamba Maisha Intervention has three key parts: A. Agricultural Commodities: KickStart "Starter Pump" (~$60 USD, 2.5 Kg), hosing, fertilizer, and seeds. B. Training: We developed model farms near each health facility where didactic and hands on training will be conducted. Our weekly didactic and practical skills training will rotate topics to ensure all participants receive full coverage. Women will be encouraged to invite a key farming support person to trainings. C. Model farm harvest: Participants will harvest vegetables at the model farms for their own consumption until their individual farms start producing in 6-8 weeks to ensure access to a nutritious diet from the time of enrollment.
  Arms: Agricultural tools and training

SUMMARY:
Scarcity of food is a leading cause of sickness and death in mothers and their newborns in sub-Saharan Africa. Use of locally acceptable agricultural interventions including provision of agricultural supplies, training and having model farms can go a long way to alleviate the ills of food scarcity among mothers and children in our region. This study is designed to learn whether an agricultural intervention might prevent food scarcity and illness among mothers and children. A total of 410 pregnant women will be enrolled from 9- 20 weeks of pregnancy, half living with HIV. Women will be randomly assigned to receive the intervention right away or to receive the intervention after the study is over if they are interested. Follow-up on enrolled participants will happen at a specified period of time, up to 12 months postpartum. The central hypothesis is that by empowering pregnant women with skills and commodities for sustainable farming, the intervention will lead to better maternal and infant health compared to control participants. The study intervention includes the provision of agricultural commodities (including irrigation pumps seeds, and other supplies) training on agriculture and business, and a demonstration farm where all trainings will be held and where women can harvest vegetables to bring home. The study aims to explore the impact of the intervention on health outcomes as well as socioeconomic and behavioral factors among the study population. This research will significantly advance scientific understanding of the importance of such agricultural interventions for pregnant women and their infants in the first year of life.

DETAILED DESCRIPTION:
Food insecurity is a critical driver of maternal and infant health and nutrition, including poor birth outcomes, suboptimal breastfeeding, perinatal depression and stress, and poor child growth and development. Pregnant women living with HIV are particularly vulnerable to food insecurity and face an excess risk of poor birth and infant outcomes. In sub-Saharan Africa, where both food insecurity and HIV are highly prevalent and a third of children under five are stunted, interventions to reduce food insecurity and malnutrition that are relevant for women with and without HIV are needed. In rural settings in this region, small-scale farming is the primary source of livelihood, yet unpredictable rainfall, severe climate events, and limited irrigation hamper crop yields. Agricultural livelihood interventions are a promising approach to raising income, bolstering food security, and ultimately improving maternal and infant health and nutrition. However, studies of agricultural interventions initiated in pregnancy are lacking despite the fact that in utero exposures crucially predict pregnancy and infant outcomes. The overall objectives of this proposal are to determine the effectiveness of an agricultural livelihood intervention on improving maternal and infant health when initiated in early pregnancy, and to understand factors that influence implementation of the agricultural intervention in the perinatal period, including the need for farming support when pregnancy impacts women's capacity to work in the field.

This is a hybrid effectiveness implementation clinical trial among 410 pregnant women enrolled at ≤from 9 -20 weeks gestation, half living with HIV in western Kenya. Women will be randomized 1:1 to the intervention or routine care. The proposed agricultural intervention package will include: a. Supply of agricultural commodities of, irrigation pump, seeds and fertilizers b. Training in agriculture, agribusiness and safety c. Model farm to enhance training and earlier harvest for food. The intervention will be implemented soon after enrolment. The study aims include: Aim 1: Determine the impact of the intervention on maternal, pregnancy and infant health outcomes. Aim 2: Determine the impact of the intervention on empowerment, socioeconomic, and behavioral factors that may influence maternal and infant health. Aim 3: Identify attitudes, norms, processes, and resources that influence implementation outcomes and effectiveness of the intervention initiated in early pregnancy. Follow up with clinical and anthropometry measures will be conducted for all the enrolled participants at 30 weeks and 36 weeks, delivery, and at 6 weeks, 3 months, 6 months, 9 months, and 12 months postpartum. The central hypothesis is that by empowering pregnant women with skills and tools for sustainable farming and perinatal nutrition, the intervention will lead to improved maternal and infant health compared to control participants. An HIV status neutral approach will optimize the generalizability and potential reach of this intervention. Also, because HIV stigma and poor health present additional barriers to empowerment and healthy behaviors, this intervention, which may reduce these barriers, has the potential to alleviate infant health disparities associated with maternal HIV.

This proposed research is highly significant because it will address a critical gap in evidence of locally effective, acceptable, feasible, adaptable and scalable interventions that may lead to improved maternal and infant nutritional needs. We anticipate that a deliberate neutral HIV status approach is the best as it will enable generalizability for community applications.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant and 9-20 weeks gestation confirmed by ultrasound
* singleton pregnancy
* Age ≥16 years
* moderate-severe household food insecurity or malnutrition (mid-upper arm circumference (MUAC) <23 cm)
* Access to land and permanent surface water
* self-reported experience with farming

Exclusion Criteria:

* Advanced HIV disease
* Unable to provide written informed consent (use of an impartial witness is satisfactory if illiterate)
* Plans to relocate outside the study area within 18 months

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 410 (Estimated)
Dates: Start 2025-09-05 (Actual); Primary Completion 2029-02-19 (Estimated); Study Completion 2029-02-19 (Estimated)

PRIMARY OUTCOMES:
Infant length for age at 12 months | 12 months of age
  z-score for length for age using the WHO Child Growth Standards
Birth Weight | Measured at birth
  Birthweight measured to nearest 10 grams with a portable digital baby scale
Household Food Insecurity Scale (HFAIS) | Baseline, 30 weeks gestation, 36 weeks gestation, 6 weeks, 3 months, 6 months, and 12 months post-partum.
  Household Food Insecurity Access Scale (HFIAS). Scores ranges from 0-27, with higher scores indicating higher food insecurity.

SECONDARY OUTCOMES:
Low Birthweight | Measured at Birth
  <2500 grams measured using a portable digital baby scale (Seca)
Preterm birth (PTB) | Measured at delivery
  Gestational age at delivery <37 weeks
Edinburgh Postnatal Depression Scale (EPDS) | Baseline, 30 weeks gestation, 36 weeks gestation, 6 weeks, 3 months, 6 months, and 12 months post-partum.
  Scores range from 0 to 30, with higher scores indicating a greater likelihood of depression.
Stunting among infants | 12 months of age
  <-2 z-score for length for age using the WHO Child Growth Standards
Sexual Relationship Power Scale (SRPS) | Baseline
  Values for Relationship Control range from 15-60 with higher scores representing higher sexual relationship power

CONTACTS AND LOCATIONS:
Overall Officials: Craig R Cohen, MD MPH, Principal Investigator — University of California, San Francisco; Pamela M Murnane, PhD MPH MLIS, Principal Investigator — University of California, San Francisco; Phelgona A Otieno, MBChB MMed MPH, Principal Investigator — Kenya Medical Research Institute
Locations (1):
- Kenya Medical Research Institute, Nairobi, Kenya

IPD SHARING:
Plan to Share IPD: No